CLINICAL TRIAL: NCT00613730
Title: Phase II, Multi-center, Open-label, Single-Arm Study Using Gemcitabine and Panitumumab in the First-line Treatment of Subjects With Locally Advanced Unresectable or Metastatic Adenocarcinoma of the Pancreas
Brief Title: Adenocarcinoma of the Pancreas Treated With Panitumumab and Gemcitabine Regimen to Investigate Overall Survival as Primary Endpoint
Acronym: APPRISE 1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: APPRISE closure prompted by SWOG S0205 not meeting primary endpoint-improving OS. APPRISE enrollment closure due to similar design;no unexpected safety data
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20060542
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2013-11

CONDITIONS: Cancer of Pancreas; Cancer of the Pancreas; Pancreas Cancer; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Panitumumab

ARMS (1):
- Gemcitabine + panitumumab (Experimental): Panitumumab 6 mg/kg was administered intravenously (IV) before gemcitabine on Day 1 of Weeks 1, 3, 5, and 7, and then every 2 weeks (day 1 and 15) of each subsequent 4-week chemotherapy cycle. Gemcitabine 1000 mg/m^2 was administered IV once weekly (on Day 1) for 7 weeks, followed by a 1-week rest period. In subsequent cycles, gemcitabine was given once weekly (on Day 1) for 3 consecutive weeks followed by 1 week of rest. Panitumumab and gemcitabine treatment continued until disease progression, unacceptable adverse events, death, or study withdrawal occurred.
  Interventions: Drug: Gemcitabine; Drug: panitumumab

INTERVENTIONS:
Drug: Gemcitabine — Intravenous administration
  Other Names: Gemzar
Drug: panitumumab — Intravenous administration

SUMMARY:
This is a phase II, multi-center, open-label, single-arm clinical trial to be conducted in the United States. In approximately 55 centers, approximately 75 eligible locally advanced unresectable or metastatic pancreatic cancer subjects will be enrolled to receive first-line therapy of gemcitabine and panitumumab.

DETAILED DESCRIPTION:
Enrollment closed after 3 patients were enrolled. This voluntary action was prompted by the announcement that the Southwest Oncology Group (SWOG) S0205 trial (NCT00075686), A Phase III Randomized Open Label Study Comparing Gemcitabine Plus Cetuximab (IMC-C225) Versus Gemcitabine as First-Line Therapy of Patients with Advanced Pancreas Cancer, did not meet its primary endpoint of improving overall survival).

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 and ≤ 75 years of age
* Histologically or cytologically confirmed pancreatic adenocarcinoma meeting one of the following criteria: Locally advanced unresectable disease, or metastatic disease
* Measurable or unmeasurable disease
* Patients with unresectable pancreatic cancer who have had surgery (exploratory laparotomy, bilary, gastrointestinal bypass) are eligible, if the patient has fully recovered from surgery and ≥ 28 days has passed since the operation. Patients with history of pancreatoduodenectomy are eligible provided that there is radiographically documented disease recurrence
* Karnofsky performance score ≥ 60 %
* Life expectancy of ≥ 12 weeks as documented by the investigator
* Hematologic function, as follows: Absolute neutrophils count (ANC) ≥ 1.5 x 10^9/L, platelet count ≥ 100 x 10^9/L, and hemoglobin ≥ 9.0 g/dL
* Renal function, as follows: Serum creatinine ≤ 1.5 mg/dL
* Hepatic function, as follows: Aspartate aminotransferase (AST) ≤ 3 x upper limit of normal (ULN) (if liver metastases ≤ 5 x ULN), alanine aminotransferase (ALT) ≤ 3 x ULN (if liver metastases ≤ 5 x ULN), and total bilirubin ≤ 2.0 mg/dL. Patients with history of biliary obstruction are eligible after intervention, once this criteria is met.
* Metabolic function, as follows: Magnesium ≥ lower limit of normal, and calcium ≥ lower limit of normal
* Competent to comprehend, sign, and date an International Ethics Committee/Institutional Review board (IEC/IRB)-approved informed consent form

Exclusion Criteria:

* Islet cell or acinar cell carcinoma or cystadenocarcinoma
* History or known presence of central nervous system (CNS) mestatases
* History of another primary cancer, except: Curatively treated cervical carcinoma in situ, or curatively resected non-melanomatous skin cancer, or other primary solid tumor curatively treated with no known active disease present and no treatment administered for ≥ 3 years prior to enrollment
* Other concurrent anticancer chemotherapy
* Concomitant malignant disease
* Prior radiotherapy ≤ 14 days, or if subjects has not recovered from radiotherapy
* Uncontrolled seizure disorder or other serious neurological diseases
* Any co-morbid disease that would increase risk of toxicity
* Prior anti-Epidermal growth factor receptor (EGFr) antibody or Vascular endothelial growth factor (VEGF) therapy (eg, cetuximab, bevacizumab) or treatment with small molecule EGFr inhibitors (eg, gefitinib, erlotinib, lapatinib)
* Adjuvant chemotherapy or chemoradiotherapy ≥ 24 weeks prior to enrollment
* Prior treatment with gemcitabine
* Patients requiring chronic use of immunosuppressive agents (eg, methotrexate, cyclosporine, corticosteroids)
* Regular use (as determined by the investigator) of nonsteroidal anti-inflammatory agents
* Known allergy to panitumumab or any components of panitumumab formulation or gemcitabine
* Recent infection requiring a course of systemic anti-infectives that was completed ≤ 14 days before enrollment (exception can be made at the judgment of the investigator for oral treatment of an uncomplicated urinary tract infection [UTI])
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year prior to enrollment
* History of interstitial lung disease (eg, pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease) on screening chest x-ray or computed tomography (CT) scan
* Pulmonary embolism, deep vein thrombosis, or other significant thromboembolic event ≤ 8 weeks prior to enrollment
* Pre-existing bleeding diathesis or coagulopathy with the exception of well-controlled chronic anticoagulation (eg, coumadin or heparin therapy). Patients receiving coumadin should have their International Normalized Ratio (INR) monitored closely
* History of any medical or psychiatric condition or addictive disorder, or laboratory abnormality that, in the opinion of the investigator, may increase the risks associated with study participation or study drug administration or may interfere with the conduct of the study or interpretation of study results
* Patient unwilling or unable to comply with study requirements
* Patient who is pregnant or breast feeding
* Man or woman of child bearing potential (women who are post menopausal < 52 weeks, not surgically sterilized, or not abstinent) who do not consent to use adequate contraceptive precautions (per institutional standard of care) during the course of the study and for 24 weeks for women and 4 weeks for men, after the last dose of gemcitabine or panitumumab, whichever dose is last
* Known positive test(s) for human immunodeficiency virus infection, hepatitis C virus, chronic active hepatitis B infection
* Major surgery ≤ 28 days or minor surgery ≤ 14 days prior to enrollment
* Documented history of alcohol, cocaine or intravenous drug abuse ≤ 6 months of enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 26 March 2007 through 13 April 2007
Period: Overall Study
Arm/Group | Gemcitabine + Panitumumab
Started | 3
Completed | 0
Not Completed | 3
Not completed — Disease progression | 2
Not completed — Administrative decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine + Panitumumab
Number analyzed (Participants) | 3
Age Continuous [Median (Full Range); unit: years] | 64 [61 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 1
  White or Caucasian | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 1 Year
Description: The survival time is calculated from Study Day
  1 (ie, the first day that a participant receives study treatment with the gemcitabine regimen in combination with panitumumab) to the date of death due to any cause.
Time Frame: 12 months
Population: Study was terminated after enrolling 3 participants. This outcome was not evaluated.
Arm/Group | Gemcitabine + Panitumumab
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression-free Survival
Description: Progression-Free Survival was defined as the time from Study Day 1 to the date of disease progression or the date of death due to any cause (whichever comes earlier). Disease progression is determined per Response Evaluation Criteria in Solid Tumors (RECIST) criteria or per physician's assessment based on symptom progression.
Time Frame: Up to 25 months
Population: Study was terminated after enrolling 3 participants. This outcome was not evaluated.
Arm/Group | Gemcitabine + Panitumumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Participants With Overall Response
Description: Overall Response defined as the percentage of participants with complete or partial response (CR or PR), as defined by modified RECIST. CR: Disappearance of all target and non-target lesions. PR: Either at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of the longest diameters (SLD) and no progression of existing non-target lesions and no new lesions, or, the disappearance of all target lesions with persistence of one or more non-target lesion(s) not qualifying for either CR or progressive disease and no new lesions.
Time Frame: Overall study
Population: Study was terminated after enrolling 3 participants. This outcome was not evaluated.
Arm/Group | Gemcitabine + Panitumumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: First dose through maximum of safety follow-up or 30 days after last dose, up to 25 months.
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Gemcitabine + Panitumumab
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine + Panitumumab (N=3)
Asthenia (General disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine + Panitumumab (N=3)
Anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Erythema of eyelid (Eye disorders) | 1
Eye disorder (Eye disorders) | 1
Retinal oedema (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Fatigue (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Bacterial sepsis (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Weight decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Amnesia (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 1
Disorientation (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Acute prerenal failure (Renal and urinary disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial resul